CLINICAL TRIAL: NCT04320030
Title: Pilot Feasibility Study: Inflammation and Presence of M2 Macrophages Explorations With[18F]-DPA-714 PET/CT in Triple Negative Breast Cancers
Brief Title: [18F]-DPA-714 PET/CT (Positron Emission Tomography/Computerized Tomography) in Triple Negative Breast Cancers
Acronym: EITHICS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Institut Cancerologie de l'Ouest (Other)
Collaborators: SIRIC ILIAD (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ICO-N-2019-04
Record Dates: First submitted 2020-02-20; First posted 2020-03-24 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2022-08

CONDITIONS: Triple Negative Breast Cancer
Keywords: [18F]-DPA-714; Positron Emission Tomography/Computerized Tomography (PET/CT) scan; 18 kDa Translocator Protein (TSPO); Macrophages M1 and M2 detection; Immunohistochemical analysis; Diffusion-weighted breast Magnetic resonance imaging (MRI); Tumor Autoradiography; Tumor molecular subtyping
MeSH Terms: conditions — Triple Negative Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Multicentric, open prospective study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- [18F]-DPA-714 (Experimental): pretherapeutic [18F]-DPA-714 PET/CT scan
  Interventions: Drug: [18F]-DPA-714 PET/CT scan

INTERVENTIONS:
Drug: [18F]-DPA-714 PET/CT scan — Pretherapeutic [18F]-DPA-714 PET/CT scan

SUMMARY:
This phase II study is assessing the correlation between M1/M2 macrophage polarization determined by tumor immunohistochemistry analysis and [18F]DPA-714 PET/CT binding (qualitative and texture analysis) in patients with operable triple negative breast cancer.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the correlation of inflammation assessed by M1/M2 macrophage polarization determined by tumor immunohistochemistry analysis and [18F] DPA-714 PET imaging by using qualitative and image texture analysis in patients with triple negative breast cancer.

Patients receive pre-therapeutic diffusion-weighted breast MRI (Magnetic resonance imaging) and 18FDG (fluorodeoxyglucose) PET/CT (Positron Emission Tomography/Computerized Tomography) scan within 30 days before enrollment.

[18F] DPA-714 PET/CT scan is performed before surgery. About 3 MBq/Kg of [18F] DPA-714 are injected intravenously, two acquisition sequences are performed following injection and 60 minutes after injection in order to evaluate early and late tumor uptake of [18F] DPA-714.

Surgery is scheduled after [18F] DPA-714 PET/CT scan. Tissue samples from breast surgery are used to assess M1 and M2 macrophages expression and to perform tumor molecular subtyping by Immunohistochemical analysis. Tumor Autoradiography with the TSPO (18 kDa Translocator Protein) ligand [18F]DPA-714 will be also assessed on tumor tissue.

A blood sample is performed before [18F] DPA-714 PET/CT scan in order to assess the genotyping of TSPO (18 kDa Translocator Protein) gene.

ELIGIBILITY:
Inclusion Criteria:

* 18 Years and older
* Triple negative primary breast cancer based on immunohistochemical results as follows:

  * Estrogen receptor < 10%
  * And Progesterone receptors < 10%
  * And HER2 (Human Epidermal Growth Factor Receptor-2) not amplified or not overexpressed
* Patient with a primary tumor eligible for primary surgery
* Performance Status equal to 0 or 1
* Fertile patients must use effective contraception
* Patient must be affiliated to a Social Health Insurance
* Written informed consent

Exclusion Criteria:

* Patient with No triple negative breast cancer
* Patient with inflammatory breast cancer
* Patient with metastatic breast cancer
* Patient receiving cancer treatments such as chemotherapy, immunotherapy, biologic response modifiers, hormonal therapy, and radiotherapy BEFORE the biopsy and PET scans are performed
* Treated diabetes with fasting blood glucose > 10 mmol/L
* Patient who received antibiotics and/or steroidal and/or non-steroidal anti-inflammatory drugs within 30 days PRIOR to [18F]-DPA-714 PET scan
* Contraindication to MRI (implants or metallic prosthesis, severe claustrophobia, pacemaker ...)
* Patient deprived of liberty, under a measure of safeguard of justice, under guardianship or under the authority of a guardian
* Pregnant or nursing patient
* Agitation; impossibility of lying motionless for at least 1 hour, or known claustrophobia

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2020-06-11 (Actual); Primary Completion 2021-07-21 (Actual); Study Completion 2021-07-21 (Actual)

PRIMARY OUTCOMES:
Correlation between M1/M2 macrophage polarization and [18F]DPA-714 PET/CT binding | 18 months
  M1/M2 macrophage polarization will be assessed by tumor immunohistochemistry analysis, [18F]DPA-714 PET/CT binding will be assessed by qualitative and images texture analysis

SECONDARY OUTCOMES:
Correlation between TSPO genotyping (HAB = High Affinity Binder, MAB = Mixed Affinity Binder and LAB = Low Affinity Binder) and [18F]DPA-714 PET/CT binding | 18 months
  A blood sample is performed before [18F] DPA-714 PET/CT scan in order to assess the genotyping of TSPO gene at the end of study
Assess the value of early and late [18F]-DPA-714 PET/CT acquisitions | 18 months
  Early and Late tumor uptake of [18F]-DPA-714 will be assessed by qualitative and quantitative parameters measurement
Evaluate the performance of the three types of imaging used in this study: [18F]-DPA-714 PET/CT (early and late), 18FDG PET/CT and diffusion-weighted breast MRI in the characterization of triple negative breast cancer | 18 months
  This evaluation will be done by image texture analyses
Perform tumor molecular subtyping | 18 months
  This tumor molecular subtyping will be performed on breast surgery tissue samples by immuno-histochemical analysis using a panel of antibodies
[18F]-DPA-714 toxicity | 18 months
  [18F]-DPA-714 toxicity will be assessed by vital signs monitoring within 2 hours after [18F]-DPA-714 injection. Body Temperature, Pulse Rate and Blood Pressure will be mesured within two hours after [18F]-DPA-714 injection. All adverse events due to [18F]-DPA-714 will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Caroline ROUSSEAU, MD, PhD, Principal Investigator — Institut de Cancerologie de l'Ouest
Locations (3):
- France (3):
  - APHP - Hôpital Tenon, Paris
  - Institut de cancerologie de l'Ouest, Saint-Herblain
  - CHU Bretonneau, Tours